CLINICAL TRIAL: NCT06084819
Title: A Prospective,Randomized,and Comparative Study on the Efficacy of Venetoclax Combined With CACAG Regimen and BAT Regimen in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Clinical Study of Venetoclax Combined With CACAG Regimen in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: 940 Hospital of the People's Liberation Army Joint Logistic Support Force (Other); The General Hospital of Western Theater Command (Other); The General Hospital of Northern Theater Command (Other); The 960th Hospital of Joint Logistics Support Force of Chinese People's Liberation Army (Unknown); Air Force Military Medical University, China (Other); Yantai Yuhuangding Hospital (Other); People's Liberation Army (PLA) Strategic Support Force Characteristic Medical Center (Unknown); First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Daihong Liu, doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S2023-413-01
Record Dates: First submitted 2023-10-10; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-02

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia
Keywords: Relapsed/Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Clinical Protocols

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Venetoclax Combined With CACAG Regimen (Experimental): Venetoclax combined with CACAG regimen for relapsed/refractory AML. Recipients were randomized and those entering the experimental group received azacytidine,cytarabine,aclacinomycin,chidamide,venetoclax and granulocyte colony-stimulating factor. Azacytidine was used as 75 mg/m2/day from day 1 to day 7.Cytarabine was used as 75-100 mg/m2 bid from day 1 to day 5. Aclacinomycin was used as 20 mg/day on days 1,3,5. Chidamide was used as 30 mg/day on days 1,4,8,11. Venetoclax was used as 400 mg/day from day 1 to day 14.Granulocyte colony-stimulating factor was used as 300 ug/day from day 0 until agranulocytosi recovery.
  Interventions: Drug: Azacytidine;Cytarabine;Aclacinomycin;Chidamide;Venetoclax;Granulocyte colony-stimulating factor
- Best-Available Therapy(BAT) Regimen (Active Comparator): BAT regimen for relapsed/refractory AML.Recipients were randomized and those entering this group received FLAG/CLAG/MAE/DCAG/HAA/HAD regimen.
  Interventions: Drug: Best-Available Therapy(BAT) Regimen

INTERVENTIONS:
Drug: Azacytidine;Cytarabine;Aclacinomycin;Chidamide;Venetoclax;Granulocyte colony-stimulating factor — 1. Azacytidine (75mg/m2/day, days 1 to 7).
  2. Cytarabine (75-100mg/m2 q12h, days 1 to 5).
  3. Aclacinomycin(20mg/day, days 1,3,5).
  4. Chidamide(30mg/day , days 1,4,8,11).
  5. Venetoclax (100mg on day 1,200mg on day 2,400mg on days 3-14).
  6. Granulocyte colony stimulating factor (300 μg/day, day 0 until agranulocytosis recovery)
  Other Names: CACAG+VEN
  Arms: Venetoclax Combined With CACAG Regimen
Drug: Best-Available Therapy(BAT) Regimen — 1. FLAG regimen:Fludarabine(30mg/m2,days 1-5)+Cytarabine (1-2g/m2 applied 4h after fludarabine, days 1 to 5)+Granulocyte colony-stimulating factor(300ug/day,days 0 to 5)
  2. CLAG regimen:Cladribine(5mg/2,days 1-5)+Cytarabine (1-2g/m2 applied 4h after fludarabine, days 1 to 5)+Granulocyte colony-stimulating factor(300ug/day,days 0 to 5)
  3. MAE regimen:Mitox(10mg/m2,days 1 to 5)+VP-16(100mg/m2,days 1 to 5)+Cytarabine (100-150mg/m2,days 1 to 7)
  4. DCAG regimen:Decitabine(20mg/m2,days 1 to 5)+Aclacinomycin(20mg/day on days 1,3,5)+Cytarabine (100mg q12h,days 1 to 5)+Granulocyte colony-stimulating factor(300 ug/day,day 0 until agranulocytosi recovery)
  5. HAA regimen:HHT(2mg/m2,days 1 to 7)+Aclacinomycin(20mg/day,days 1 to 7) and Cytarabine (100-200 mg/m2, days 1 to 5);
  6. HAD regimen:HHT(2mg/m2,days 1 to 7)+Daunorubicin(45mg/m2/day,days 1 to 3)+Cytarabine (100-200 mg/m2,days 1 to 5).
  Other Names: FLAG/CLAG/MAE/DCAG/HAA/HAD Regimen
  Arms: Best-Available Therapy(BAT) Regimen

SUMMARY:
The purpose of this study is to compare the efficacy and safety of venetoclax combined with CACAG regimen with BAT regimen in the treatment of relapsed/refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
Despite advances in therapies for acute myeloid leukemia (AML) in the past decades, some patients still suffer from relapsed/refractory (R/R) disease, resulting in poor outcomes. With a median overall survival (OS) of 4-7 months under classic chemotherapy approaches, it is imperative to explore new treatment options.Accumulating research has demonstrated the importance of epigenetic modification in the pathogenesis of chemoresistance. Recent studies have shown that combining venetoclax with hypomethylating agents (HMAs) such as azacitidine, or low-dose cytarabine (LDAC) improves the response and survival rates in R/R AML patients. To enhance the response rate, we designed a regimen that combines chidamide, azacitidine, cytarabine, aclarubicin, and G-CSF with venetoclax (CACAG+VEN regimen) for the treatment of patients with R/R AML. In this study, we intend to compare the efficacy and safety of venetoclax combined with the CACAG regimen with Best-Available Therapy(BAT) regimen in the treatment of relapsed/refractory acute myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to understand and willing to sign the informed consent form (ICF).
* All patients should aged 14 to 75 years,no gender limitation.
* Patients with R/R AML, diagnosed in accordance with the 2021 edition of the CMA criteria
* Liver function: ALT and AST≤2.5 times the upper limit of normal ,bilirubin≤2 times the upper limit of normal;
* Renal function: creatinine ≤the upper limit of normal;
* Patients without any uncontrolled infections , without organ dysfunction or without severe mental illness;
* The score of Eastern Cooperative Oncology Group (ECOG) is 0-3,and the predicted survival ≥ 4 months.
* Patients without severe allergic constitution.

Exclusion Criteria:

* Patients with allergy or contraindication to the study drug;
* Female patients who are pregnant or breast-feeding.
* Patients with a known history of alcohol or drug addiction on the basis that there could be a higher risk of non-compliance to study treatment;
* Patients with mental illness or other states unable to comply with the protocol;
* Less than 6 weeks after surgical operation of important organs.
* Liver function: ALT and AST>2.5 times the upper limit of normal ,bilirubin>2 times the upper limit of normal;Renal function: creatinine >the upper limit of normal;
* The patient is not suitable for this clinical trial (poor compliance, substance abuse, etc.)

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) after 1 course of treatment | 1 months after the start of study treatment
  Defined as the percentage of participants achieving a best overall response of complete response (CR), CR with incomplete blood count recovery (CRi), or partial response (PR).Biological characteristics exploratory studies were analyzed by single-cell sequencing and Atac-seq. Further, according to European LeukemiaNet risk group, we analyzed the outcomes of patients by molecular subtype as a sub-group analysis.

SECONDARY OUTCOMES:
Complete Remission (CR) Rate after 1 course of treatment | 2 months after study treatment
  Defined in accordance with the IWG Response Criteria in AML. Bone marrow blasts<5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions.
Complete Remission (CR) Rate after 2 courses of treatment | After two courses of chemotherapy (each course is 28 days)
  Defined in accordance with the IWG Response Criteria in AML. Bone marrow blasts<5 percent; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L (1000/µL); platelet count >100 x 109/L (100,000/µL); independence of red cell transfusions.
Overall Response Rate (ORR) after 2 course of treatment | After two courses of chemotherapy (each course is 28 days)
  Defined as the percentage of participants achieving a best overall response of complete response (CR), CR with incomplete blood count recovery (CRi), or partial response (PR).Biological characteristics exploratory studies were analyzed by single-cell sequencing and Atac-seq. Further, according to European LeukemiaNet risk group, we analyzed the outcomes of patients by molecular subtype as a sub-group analysis.
Rate of Minimal Residual Disease (MRD)-Negative Response | After two courses of chemotherapy (each course is 28 days)
  Percentage of participants who achieved MRD-negative response, defined as < 1 leukemia cell per 10,000 leukocytes as assessed by flow cytometry.
Event-free survival | 180 days after study treatment
  Defined as the time interval from treatment initiation to the occurrence of induction failure,relapse,or death,whichever came first.
Overall Survival (OS) | 180 days after study treatment
  Defined as the time from joining the clinical study to death due to any cause.
Treatment-related adverse events | From the first dose of study treatment to 30 days after the discontinuation of treatment
  Defined as adverse events that occurred from the first dose of study treatment to 30 days after the discontinuation of treatment.
Early death | Within 30 days of the start of the first course of treatment
  Defined as death within 30 days of chemotherapy.
Disease-free survival | 180 days after study treatment
  Defined as the time interval from disease remission to the occurrence of relapse or death,whichever came first.

CONTACTS AND LOCATIONS:
Overall Officials: Daihong Liu, doctor, Study Chair — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China